CLINICAL TRIAL: NCT01793025
Title: Adoptive Transfer of Alloreactive Cells to Treat Patients With Poor-Prognosis Acute Myeloid Leukemia-01
Brief Title: Mismatched Donor Cells to Treat Acute Myeloid Leukemia
Acronym: ATAC-AML-01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Krakow, Fellow, Hematopoietic Cell Transplantation, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATAC-AML-01
Record Dates: First submitted 2013-02-10; First posted 2013-02-15 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: leukemia; myeloid; acute; acute myeloid leukemia; allogeneic; transient chimerism; cell therapy; immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

ARMS (1):
- ATAC Therapy (Experimental)
  Interventions: Biological: ATAC Therapy

INTERVENTIONS:
Biological: ATAC Therapy — Unselected peripheral blood mononuclear cells given 24-48 hours after induction or consolidation chemotherapy
  Other Names: Unselected Peripheral Blood Mononuclear Cells

SUMMARY:
The purpose of this study is to assess the safety and efficacy of infusing immune cells from a donor as treatment for patients with acute myeloid leukemia that is resistant to chemotherapy or who have experienced relapse. Unlike standard bone marrow or stem cell transplantation which uses donors who are well 'matched' to the patient, this study uses donors whose immune cells are not compatible with the patient. With standard stem cell or bone marrow transplantation, the well-matched immune cells will attack the leukemia but they also attack the patient's organs (a situation called graft-versus-host disease, which can persist in the long term). Our hypothesis is that the mismatched donor cells will fight the leukemia but will then be eliminated from the patient's body, so long-term side effects like graft-versus-host disease should not occur.

DETAILED DESCRIPTION:
The ATAC cell therapy product contains unselected, non-mobilized peripheral blood mononuclear cells from related donors who are mismatched to the recipients at 3 or more (out of 6) HLA loci. Cohorts of 3 patients will be treated at each of four pre-specified dose levels (T cells per kg recipient weight). One ATAC infusion is administered 24-48 hours following re-induction chemotherapy (for relapsed or primary refractory AML patients not in remission). In situations where ATAC infusion is not available immediately following re-induction chemotherapy and patients nonetheless achieve complete remission, one ATAC infusion is given 24-48 hours after consolidation chemotherapy.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Age ≥ 18 years (no upper age limit, but physician discretion is advised)
* AML that is refractory to 2 courses of induction therapy (that together constitute the 'first-line' therapy) or that has relapsed after a period of morphologic complete remission or morphologic remission with incomplete blood count recovery (CRi)
* Candidacy for intense induction chemotherapy (ECOG 0-2, adequate renal, liver and cardiac function, absence of uncontrolled infections)
* Availability of parents, siblings or children who are HLA haploidentical (and not homozygous for the shared haplotype), who are deemed suitable donors after medical evaluation, and who complete peripheral blood mononuclear cell collection
* No history of autologous or allogeneic stem cell transplant, purine analog chemotherapy or cyclophosphamide, or total body irradiation
* Ability to comprehend the investigational nature of the study and provide informed consent

Recipient Exclusion Criteria:

* Acute promyelocytic leukemia (including those with non-classical rearrangements of RARα)
* History of severe myelodysplastic syndrome clearly preceding the diagnosis of AML (i.e., red cell transfusion dependence or erythropoietin dependence over a 4-month period, or in the absence of a clear cause, any of the following: hemoglobin consistently below 9 g/dL or platelets below 50 x 10^9/L or ANC below 1000/uL on 2 or more occasions 2 weeks apart, or use of G-CSF to maintain the ANC threshold in the absence of infection, in the 3 months preceding the diagnosis of AML). Exception: If ATAC therapy is being considered as a bridge to stem cell transplantation in patients with an available standard transplant donor (familial, unrelated, or cord blood), this exclusion criterion does not apply.
* Grade 2-3/3 fibrosis in the diagnostic bone marrow biopsy
* DLCO < 40% predicted
* Left ventricular ejection fraction < 40% (evaluated by ECHO or MUGA)
* AST/SGOT > 2.5 x ULN
* Bilirubin > 1.5 x ULN
* Creatinine > 1.5 x ULN
* Creatinine clearance < 50 mL/min
* HIV positive
* Major anticipated illness or organ failure incompatible with survival from chemotherapy
* Concurrent second primary cancer or a prior malignancy that required cytotoxic treatment within the past 12 months, other than cervical carcinoma in-situ or prostate cancer in-situ
* Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the treatment unlikely and informed consent impossible
* Any congenital or acquired immunodeficiency that would possibly permit permanent engraftment of donor cells
* Receiving systemic steroid therapy or systemic immunosuppression such as cyclosporine or TNF-inhibitors
* Prior or concurrent receipt of any marketed or investigational agent deemed on an ad hoc basis to cause immunomodulation, pose a threat of permanent engraftment or increase the risk of GVHD.

Donor inclusion criteria:

* Mismatched family donor (incompatibility at 3 loci HLA-A, B and DR of the unshared haplotype, or higher-order incompatibility)
* Age ≥ 16 and ≤ 80 years
* Fit to undergo apheresis (normal blood counts, normotensive and no history of stroke).
* Donor has been tested negative for HIV-1, HIV-2, hepatitis B virus (HBV, surface and core antigen), hepatitis C virus, human T-lymphotropic virus types I/II, and Treponema pallidum (syphilis).
* ECOG performance status of 2 or less.
* Adequate veins for leukapheresis or agree to placement of a temporary central venous catheter.
* Donor must provide written informed consent.
* Where multiple equally-suitable donors are available, sex mismatched donors will be preferred.

Donor exclusion criteria:

* Medically uncontrolled coronary heart disease
* Myocardial infarction within the last 3 months
* History of seizure
* History of stroke
* History of malignancy (except basal cell or squamous carcinoma of the skin, or positive PAP smear and subsequent negative follow-up)
* Presence of a transmissible disease (such as HIV seropositivity)
* Presence of a major illness or a suspected systemic dysfunction
* Presence of an an active inflammatory or autoimmune disorder
* Female donors who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Safety | 60 days (up to 2 years)
  Maximum tolerated cell dose: Dose at which < 33% of patients experienced dose-limiting toxicity. If no DLT occurs, then dose titration will stop at a pre-specified number of T cells/kg. Four dose-level cohorts are planned.

SECONDARY OUTCOMES:
Treatment-related mortality | Continuous up to 2 years
Non-relapse mortality | Continuous up to 2 years
Incidence of graft-versus-host disease | Continuous up to 2 years
Duration of cytopenias | Monitored continuously from ATAC infusion until peripheral blood count recovery or maximum 2 years (whichever is earlier)
Overall survival | Continuous up to 2 years
Complete and incomplete remissions (CR, CRi) | Day 60 post cell infusion
Relapse-free survival | Continuous up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Delisle, MD,PhD, Study Chair — Hôpital Maisonneuve-Rosemont and Université de Montréal; Elizabeth Krakow, MD, Principal Investigator — Hôpital Maisonneuve-Rosemont and Université de Montréal
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada